CLINICAL TRIAL: NCT04579770
Title: Effect of Oral Ketone and Sodium Bicarbonate Administration on Physiological and Metabolic Parameters During Endurance Exercise in Hypoxia
Brief Title: Effect of Oral Ketone and Sodium Bicarbonate Administration During Endurance Exercise in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jozef Stefan Institute (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Tadej Debevec, Principal Investigator, Jozef Stefan Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: J5-9350
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Exercise; Hypoxia
Keywords: exercise; hypoxia; ketone
MeSH Terms: conditions — Motor Activity; Hypoxia; Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Only carbohydrates will be provided
  Interventions: Other: Placebo
- Ketone ester (Experimental): Ketone ester with carbohydrates will be provided
  Interventions: Dietary Supplement: Ketone ester
- Ketone ester + bicarbonate (Experimental): Ketone ester with bicarbonate and carbohydrates will be provided
  Interventions: Dietary Supplement: Ketone ester; Other: Sodium bicarbonate
- Bicarbonate (Experimental): Bicarbonate and carbohydrates will be provided
  Interventions: Other: Sodium bicarbonate

INTERVENTIONS:
Dietary Supplement: Ketone ester — 75g ketone ester in the form of a drink [96% (R)-3-hydroxybutyl (R)-3-hydroxybutyrate, Oxfordshire, UK)] will be provided.
  Arms: Ketone ester; Ketone ester + bicarbonate
Other: Sodium bicarbonate — Sodium bicarbonate - widely accessible food ingredient will be provided.
  Arms: Bicarbonate; Ketone ester + bicarbonate
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is investigating the effects of oral ketone and sodium bicarbonate administration on physiological and metabolic parameters during cycling endurance exercise in hypoxia. Ketone body supplementation is commonly used among elite endurance athletes that also compete in the hypoxia (at altitude). To-date effects of ketones have only been investigated in normoxia and the data in hypoxia is lacking. Hence, we want to investigate the effect of oral ketone ester intake with and without additional sodium bicarbonate (NaHCO3) ingestion on i) blood-acid base balance and ii) exercise performance during prolonged exercise under hypoxic conditions. Information obtained via this study should provide valuable information with regard to optimisation of exercise training and athletic performance, and more importantly, provide pioneering insight on the metabolic and physiological responses to ketosis under hypoxic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 35 years old
* Recreational or competitive cyclist performing regularly cycling training sessions of at least 4 hours, with an average training volume of more than 6 hours per week
* Good health status confirmed by a medical screening
* VO2max higher than 55 ml.min-1.kg-1
* Body Mass Index (BMI) between 18 and 25

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform high-intensity exercise
* Intake of any medication or nutritional supplement that is known to affect exercise performance
* Intake of analgesics, anti-inflammatory agents, or supplementary anti-oxidants, from 2 weeks prior to the start of the study.
* Blood donation within 3 months prior to the start of the study
* Smoking
* More than 3 alcoholic beverages per day, including a maximum of one glass of wine per day
* Involvement in elite athletic training at a semi-professional or professional level
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Cycling performance - Simulated 15-min long time trial | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Performance (average power output) during the 15 min long time trial on an ergometer
Change in Cycling performance - Simulated Sprint | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Time to exhaustion at 175% of the intensity of the second lactate threshold
Change in Blood acid-base balance (pH and [HCO3-]) during cycling | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Blood acid-base balance assement

SECONDARY OUTCOMES:
Change in Blood ketone concentrations during exercise | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Blood ketone assesment
Change in Blood glucose concentrations during exercise | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Blood glucose assesment
Change in Blood lactate concentrations during exercise | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Blood lactate assesment
Change in Respiratory parameters (VE, V̇O2 and V̇CO2) during exercise | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Gas exchange measurement
Change in arterial oxygen saturation during exercise | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Pulse oxymetry measurement
Change in muscle oxygenation during exercise | 5 hours - this is how long each experimental session is going to last. Subjects would be asked to do it 3 times as there are 3 different experimental conditions
  Near infrared spectroscopy measuremet

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium